CLINICAL TRIAL: NCT01851720
Title: Randomized Trial for Pain Management in Low-grade Subarachnoid Hemorrhage
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inclusion criteria were too strict and therefore we were not able to recruit more patients.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00071159
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Headaches Associated With Subarachnoid Hemorrhage (SAH)

ARMS (2):
- Control group / Standard of Care (Active Comparator): * IV fentanyl bolus 25-50 mcg every 1-2 hrs as needed for pain
  * (Bolus dose can be titrated up in 25 mcg increments if necessary)
  * Maximum dose of 100 mcg/hr
  Interventions: Drug: Standard IV fentanyl bolus
- Low dose IV fentanyl PCA (Active Comparator): * Initially: 10 mcg demand dose every 12 minutes
  * No initial bolus and no continuous infusion
  * Demand dose increased 10 mcg every 12 minutes if necessary
  * Maximum dose of 100 mcg/hr
  Interventions: Drug: Low dose fentanyl PCA

INTERVENTIONS:
Drug: Low dose fentanyl PCA
  Arms: Low dose IV fentanyl PCA
Drug: Standard IV fentanyl bolus
  Arms: Control group / Standard of Care

SUMMARY:
Headaches associated with subarachnoid hemorrhage (SAH) cause severe pain. Headache management is complex, requiring a balance between pain control and preservation of neurological assessment. Sufficient pain control can be achieved with narcotics, however, these carry numerous undesirable side effects. Most critically, all narcotics can result in respiratory depression and sedation. For patients who present without neurological defects but debilitating pain, management is particularly challenging. The sedative effect of narcotics confounds the management of these patients by interfering with the neurological examination. Pain management is also a significant concern for patient's families as they observe suffering without full understanding of the importance of preserved mental status. In order to control the pain associated with SAH headaches, the use of narcotics is often required despite the risks. This standard therapy involves an IV bolus dose delivered by the provider regularly as needed for pain control. A common approach to reduce pain in other patient populations, including acute pain relief following major spine surgery, is patient controlled analgesia (PCA). With the PCA method, patients deliver low doses of narcotics through a pain pump with preset maximal doses and frequency of delivery. We hypothesize that this approach to pain relief for SAH headaches will result in lower pain scores, greater patient and family satisfaction scores, and increased patient safety with lower narcotic doses minimally interfering with neurological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age>18-75
* Glasgow Coma Scale (GCS) 13 or greater
* Hunt and Hess grade I, II conditions
* Admitted within 2 days of initial SAH event >6/10 pain on presentation

Exclusion Criteria:

* Aphasia
* Head trauma within the past 30 days
* Need for craniotomy
* h/o obstructive sleep apnea or respiratory disease
* h/o opioid tolerance
* evidence of vasospasm
* h/o liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group / Standard of Care: * IV fentanyl bolus 25-50 mcg every 1-2 hrs as needed for pain
  * (Bolus dose can be titrated up in 25 mcg increments if necessary)
  * Maximum dose of 100 mcg/hr
  Standard IV fentanyl bolus
- Low Dose IV Fentanyl Patient Controlled Analgesia (PCA): * Initially: 10 mcg demand dose every 12 minutes
  * No initial bolus and no continuous infusion
  * Demand dose increased 10 mcg every 12 minutes if necessary
  * Maximum dose of 100 mcg/hr
  Low dose fentanyl PCA
Period: Overall Study
Arm/Group | Control Group / Standard of Care | Low Dose IV Fentanyl Patient Controlled Analgesia (PCA)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Dose IV Fentanyl PCA: * Initially: 10 mcg demand dose every 12 minutes
  * No initial bolus and no continuous infusion
  * Demand dose increased 10 mcg every 12 minutes if necessary
  * Maximum dose of 100 mcg/hr
  Low dose fentanyl PCA
- Total: Total of all reporting groups
Arm/Group | Control Group / Standard of Care | Low Dose IV Fentanyl PCA | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian |  | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Acute Pain Following Sub-Arachnoid Hemorrhage (SAH) is the Primary Outcome Variable and Will be Assessed Using the Numeric Rating Scale (NRS).
Description: Pain score 0-10. 0 represented no pain and 10 worst pain
Time Frame: 4 days
Population: Though one subject in the PCA arm completed enrollment, we had insufficient data to perform any comparative analysis. We do no intend to summarize the patient's results.
Arm/Group | Control Group / Standard of Care | Low Dose IV Fentanyl PCA
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Group / Standard of Care | Low Dose IV Fentanyl PCA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes